CLINICAL TRIAL: NCT00439231
Title: A Phase II Study of Lenalidomide Revlimid(Registered Trademark) in Previously Treated Patients With Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Brief Title: Lenalidomide in Previously Treated Patients With Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Georg Aue, M.D. (NIH)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Georg Aue, M.D., NHLBI Hematolgy Clinician, National Heart, Lung, and Blood Institute (NHLBI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 070104; 07-H-0104 (Other: NIH NHLBI); NCT00465127 (obsolete NCT alias)
Record Dates: First submitted 2007-02-22; First posted 2007-02-23 (Estimated); Results first posted 2014-01-13 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2013-11

CONDITIONS: Chronic Lymphocytic Leukemia (CLL); Small Lymphocytic Lymphoma
Keywords: Monoclonal Antibody Therapy; Biologic Response Modifier Therapy; CLL; SLL; chemo-care (CC) 5013- Revlimid; Chronic Lymphocytic Leukemia; Small Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide (Revlimid) subjects (Experimental): Lenalidomide regimen testing to determine efficacy for CLL/ SLL subjects
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — Lenalidomide (Revlimid) regimen testing to determine efficacy for SLL/ CLL subjects
  Other Names: Revlimid

SUMMARY:
This study will evaluate the safety and effectiveness of a new drug called lenalidomide (Revlimid) for treating patients with chronic lymphocytic leukemia (CLL) and small lymphocytic lymphoma (SLL) who relapsed after their initial treatment.

Patients 21 years of age and older with CLL or SLL who have previously received standard treatment may be eligible for this study.

Participants take lenalidomide capsules once a day for 21 days, followed by 21 days off the drug. This constitutes one treatment cycle. Treatment continues for four cycles as long as the medicine is tolerated. After four cycles, patients who respond completely continue treatment for another two cycles; patients who respond partially continue treatment for another four cycles; and patients who do not respond stop treatment but continue to be followed for safety.

...

DETAILED DESCRIPTION:
There is evidence that lenalidomide has single agent activity in chronic lymphocytic leukemia (CLL)/small lymphocytic leukemia (SLL). Optimal dosing of lenalidomide in CLL has not been established yet. A pilot clinical trial in CLL studied single agent lenalidomide cycled every 4 weeks with 25 mg for three weeks on and one week off drug. In this trial dose reductions have been necessary secondary to prolonged neutropenia or thrombocytopenia in a majority of patients. However, there was also remarkable efficacy and evidence for an immune stimulatory effect of lenalidomide. Therefore, we propose this phase II trial using 20 mg lenalidomide (Revlimid(Registered Trademark)) 3 weeks on and 3 weeks off for 4 cycles in subjects who have been previously treated for chronic lymphocytic leukemia (CLL)/small lymphocytic leukemia (SLL). Subjects with at least partial response (PR) may go on to receive 4 additional cycles.

The primary objective of the trial is to test the efficacy of a more tolerable dosing scheme of lenalidomide.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Diagnosed with chronic lymphocytic leukemia (CLL) or small lymphocytic leukemia (SLL).
  2. Failed prior standard of care therapy for CLL.
  3. Neutrophil count (ANC) greater than or equal to 500/microliter (mcL).
  4. Platelet count greater than or equal to 20,000/mcL.
  5. Age 21-99.

EXCLUSION CRITERIA:

1. Chronic or current clinically significant infection, including HIV positivity or uncontrolled infection.
2. Eastern Cooperative Oncology Group (ECOG) performance greater than 2.
3. Other concurrent anticancer therapies.
4. Less than 4 weeks from last systemic therapy for CLL. Steroids up to 2 weeks before the start of treatment are permissible.
5. Moribund status or concurrent hepatic, renal, cardiac, neurologic, pulmonary, infectious, or metabolic disease of such severity that it would preclude the patient's ability to tolerate protocol therapy.
6. Creatinine greater than 1.5 times the upper limit of normal.
7. Women who are pregnant or nursing, as well as women of childbearing potential who are unwilling to use a dual method of contraception.
8. Men who are unwilling to use a barrier protection.
9. Inability to understand the investigational nature of the study; inability to provide informed consent.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2007-02; Primary Completion 2010-09 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Georg Aue, MD, Principal Investigator — NIH National Heart, Lung, and Blood Institute
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Aue G, Nelson Lozier J, Tian X, Cullinane AM, Soto S, Samsel L, McCoy P, Wiestner A. Inflammation, TNFalpha and endothelial dysfunction link lenalidomide to venous thrombosis in chronic lymphocytic leukemia. Am J Hematol. 2011 Oct;86(10):835-40. doi: 10.1002/ajh.22114. Epub 2011 Aug 2. PMID 21812019
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2007-H-0104.html

RESULTS

PARTICIPANT FLOW:
Groups:
- CLL Subjects Response to Lenalidomide (Revlimid): To establish a response rate to lenalidomide (Revlimid) in subjects with CLL/SLL using a 3 week on, 3 week off dosing regimen. The responses will be categorized using the revised 1996 National Cancer Institute - sponsored working guidelines. The response rate will be based on changes in peripheral blood measures (ANC, platelets and/or hemoglobin), lymphadenopathy, hepatomegaly, splenomegaly or constitutional symptoms; and bone marrow biopsy measured at 24 weeks after the first dose of lenalidomide using the protocol dosing regimen. Complete responders will respond to treatment after 2 cycles. Partial responders will respond to treatment after 4 cycles.
Period: Overall Study
Arm/Group | CLL Subjects Response to Lenalidomide (Revlimid)
Started | 33
Completed | 5 (5 subjects had a partial response, 0 complete response, 28 completed off study,)
Not Completed | 28
Not completed — Lack of Efficacy | 28

BASELINE CHARACTERISTICS:
Groups:
- CLL Subjects Response to Lenalidomide (Revlimid): To establish a response rate to lenalidomide (Revlimid) in subjects with chronic lymphocytic leukemia (CLL)/ small lymphocytic leukemia (SLL) using a 3 week on, 3 week off dosing regimen. The responses will be categorized using the revised 1996 National Cancer Institute - sponsored working guidelines. The response rate will be based on changes in peripheral blood measures (ANC, platelets and/or hemoglobin), lymphadenopathy, hepatomegaly, splenomegaly or constitutional symptoms; and bone marrow biopsy measured at 24 weeks after the first dose of lenalidomide using the protocol dosing regimen. Complete responders will respond to treatment after 2 cycles. Partial responders will respond to treatment after 4 cycles.
Arm/Group | CLL Subjects Response to Lenalidomide (Revlimid)
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 26
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: To Establish the Overall Response Rate Measured at 24 Weeks After First Dose of Lenalidomide Using This Dosing Regimen
Description: To establish the overall response rate based on peripheral blood measures (absolute neutrophil count, platelets, and/or hemoglobin), lymphadenopathy, hepatomegaly, splenomegaly or constitutional symptoms; and bone marrow biopsy measured at 24 weeks after first dose of lenalidomide using this dosing regimen
Time Frame: 24 weeks of lenalidomide therapy
Measure: Number; unit: participants
Groups:
- CLL Subject Response Rate After Lenalidomide Therapy: To establish a response rate to lenalidomide (Revlimid) in subjects with chronic lymphocytic leukemia (CLL)/ small lymphocytic lymphoma (SLL) using a 3 week on, 3 week off dosing regimen. Complete responders will respond to treatment after 2 cycles. Partial responders will respond to treatment after 4 cycles.
Arm/Group | CLL Subject Response Rate After Lenalidomide Therapy
Number analyzed (Participants) | 33
participants
  Complete response | 0
  Partial response | 5
  No response | 28

ADVERSE EVENTS:
Arm/Group | CLL Subjects Treated With Lenalidomide (Revlimid)
Serious Adverse Events (participants affected / at risk) | 8/33
Other Adverse Events (participants affected / at risk) | 32/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CLL Subjects Treated With Lenalidomide (Revlimid) (N=33)
DVT (Blood and lymphatic system disorders) | 1
Tumor flare syndrome (Blood and lymphatic system disorders) | 7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CLL Subjects Treated With Lenalidomide (Revlimid) (N=33)
ankle edema (Blood and lymphatic system disorders) | 1
bruising inner arm (Blood and lymphatic system disorders) | 1
decrease in hemoglobin (Blood and lymphatic system disorders) | 8
decrease in neutrophils (Blood and lymphatic system disorders) | 19
decrease in platelets (Blood and lymphatic system disorders) | 19
DVT leg (Blood and lymphatic system disorders) | 1
elbow bruising (Blood and lymphatic system disorders) | 1
flu like symptoms (Blood and lymphatic system disorders) | 3
hematoma (Blood and lymphatic system disorders) | 2
hypophosphatemia (Blood and lymphatic system disorders) | 1
increase ALT (Blood and lymphatic system disorders) | 1
lymph node swelling (Blood and lymphatic system disorders) | 3
lymphedema (Blood and lymphatic system disorders) | 1
swollen lymph node (Blood and lymphatic system disorders) | 1
Tumor flare syndrome (Blood and lymphatic system disorders) | 13
hypotension (Cardiac disorders) | 2
decreased hearing (Ear and labyrinth disorders) | 1
ear pressure (Ear and labyrinth disorders) | 1
middle ear pain (Ear and labyrinth disorders) | 1
blurred vision (Eye disorders) | 1
dry eye (Eye disorders) | 1
edema ocular (Eye disorders) | 1
uvietus (Eye disorders) | 1
abdominal bloating (Gastrointestinal disorders) | 3
abdominal cramps (Gastrointestinal disorders) | 3
abdominal distention (Gastrointestinal disorders) | 2
abdominal pain (Gastrointestinal disorders) | 8
change in taste (Gastrointestinal disorders) | 3
constipation (Gastrointestinal disorders) | 8
decrease in creatinine (Gastrointestinal disorders) | 1
diarrhea (Gastrointestinal disorders) | 9
dry mouth (Gastrointestinal disorders) | 1
heartburn (Gastrointestinal disorders) | 1
increase ALT (Gastrointestinal disorders) | 2
increase AST (Gastrointestinal disorders) | 2
nausea (Gastrointestinal disorders) | 5
organomegaly (Gastrointestinal disorders) | 1
stomach pain (Gastrointestinal disorders) | 1
urinary tract infection (Gastrointestinal disorders) | 1
vomiting (Gastrointestinal disorders) | 3
ankle swelling (General disorders) | 1
chills (General disorders) | 4
cold sore (General disorders) | 1
cough (General disorders) | 1
fatigue (General disorders) | 19
fever (General disorders) | 5
insomnia (General disorders) | 1
lower extremity edema (General disorders) | 1
mouth lesion (General disorders) | 1
mouth/lip sore (General disorders) | 1
pedal edema (General disorders) | 1
sweating (General disorders) | 6
weight loss (General disorders) | 9
CMV infection (Infections and infestations) | 1
Gastrointestinal infection (Infections and infestations) | 1
gum infection (Infections and infestations) | 1
oral cavity infeciton (Infections and infestations) | 1
oral ulcers (Infections and infestations) | 1
shingles (Infections and infestations) | 1
tooth abscess (Infections and infestations) | 1
upper respiratory infection (Infections and infestations) | 1
arm pain (Musculoskeletal and connective tissue disorders) | 2
back pain (Musculoskeletal and connective tissue disorders) | 5
bruising arms & back (Musculoskeletal and connective tissue disorders) | 1
chest pain (Musculoskeletal and connective tissue disorders) | 1
elbow pain (Musculoskeletal and connective tissue disorders) | 2
feet pain (Musculoskeletal and connective tissue disorders) | 1
foot cramps (Musculoskeletal and connective tissue disorders) | 1
foot/ankle pain (Musculoskeletal and connective tissue disorders) | 1
general body aches (Musculoskeletal and connective tissue disorders) | 1
generalize bruising (Musculoskeletal and connective tissue disorders) | 1
hand cramps (Musculoskeletal and connective tissue disorders) | 1
joint pain (Musculoskeletal and connective tissue disorders) | 1
leg cramp (Musculoskeletal and connective tissue disorders) | 1
leg cramps (Musculoskeletal and connective tissue disorders) | 1
leg pain (Musculoskeletal and connective tissue disorders) | 2
lower extremity cramps (Musculoskeletal and connective tissue disorders) | 1
lower extremity leg cramps (Musculoskeletal and connective tissue disorders) | 1
lower extremity pain (Musculoskeletal and connective tissue disorders) | 3
lower extremity rash (Musculoskeletal and connective tissue disorders) | 1
muscle cramp (Musculoskeletal and connective tissue disorders) | 1
muscle cramps (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
neck pain (Musculoskeletal and connective tissue disorders) | 2
ocular infection (Musculoskeletal and connective tissue disorders) | 1
petechiae legs (Musculoskeletal and connective tissue disorders) | 1
pleuritic back pain (Musculoskeletal and connective tissue disorders) | 1
scalp rash (Musculoskeletal and connective tissue disorders) | 1
shoulder pain (Musculoskeletal and connective tissue disorders) | 3
skin rash (Musculoskeletal and connective tissue disorders) | 1
agitation (Nervous system disorders) | 1
hallucinations (Nervous system disorders) | 1
head/ arm nueropathy (Nervous system disorders) | 1
headache (Nervous system disorders) | 6
insomnia (Nervous system disorders) | 2
syncope (Nervous system disorders) | 12
depressed (Psychiatric disorders) | 1
upper respiratory infection (Reproductive system and breast disorders) | 1
bronchitis (Respiratory, thoracic and mediastinal disorders) | 1
cough (Respiratory, thoracic and mediastinal disorders) | 3
dyspnea (Respiratory, thoracic and mediastinal disorders) | 10
mouth lesion (Respiratory, thoracic and mediastinal disorders) | 1
pulmonary infiltrate (Respiratory, thoracic and mediastinal disorders) | 1
rales (Respiratory, thoracic and mediastinal disorders) | 1
sinus infection (Respiratory, thoracic and mediastinal disorders) | 1
sore throat (Respiratory, thoracic and mediastinal disorders) | 2
throat pain (Respiratory, thoracic and mediastinal disorders) | 1
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 16
facial rash (Skin and subcutaneous tissue disorders) | 1
hand rash (Skin and subcutaneous tissue disorders) | 1
head rash (Skin and subcutaneous tissue disorders) | 1
knee rash (Skin and subcutaneous tissue disorders) | 1
pruritis (Skin and subcutaneous tissue disorders) | 5
rash axilla (Skin and subcutaneous tissue disorders) | 1
rash chest (Skin and subcutaneous tissue disorders) | 1
rash leg (Skin and subcutaneous tissue disorders) | 1
rash scalp (Skin and subcutaneous tissue disorders) | 2
rash torso (Skin and subcutaneous tissue disorders) | 1
rash waistband (Skin and subcutaneous tissue disorders) | 1
scalp rash (Skin and subcutaneous tissue disorders) | 2
skin rash (Skin and subcutaneous tissue disorders) | 14
skin rash lip (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes